CLINICAL TRIAL: NCT00488501
Title: Clinical Usefulness and Efficacy of Intrathoracic Impedance Monitoring Using the OptiVol Patient Alert(TM) in Medtronic(R) ICD's for Early Detection of Decompensated Heart Failure
Brief Title: Clinical Usefulness and Efficacy of Intrathoracic Impedance Monitoring Using the OptiVol Patient Alert(TM)
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Mrs. A. van Pol-Spiering, Stichting Toegepast Wetenschappelijk Cardiologisch Onderzoek
Other Study IDs: M06-16106
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Heart Failure
Keywords: intrathoracic impedance; cardiac resynchronization therapy; heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study we investigate the clinical value and efficacy of OptiVol (TM) impedance measurements by Medtronic (R) ICD's. We aim to determine sensitivity and positive predictive value for detecting heart failure. We also investigate if left ventricular filling pattern measured by echocardiography and/or brain natriuretic peptide (BNP) level can be used to improve the positive predictive value of the Optivol alert

DETAILED DESCRIPTION:
Patients who have a Medtronic (R) ICD equipped with the Optivol (TM) impedance monitoring will be included in your study after informed consent. The OptiVol (TM) feature will be activated and at baseline data is collected (blood sample including BNP, electrocardiography, echocardiography, chest X-ray and ICD check-up). During follow-up patients will be re-assessed in case of an OptiVol alert or in case of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure of any cause
* implanted Medtronic ICD with OptiVol impedance monitoring

Exclusion Criteria:

* inability to receive informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have been implanted a biventricular pacemaker ICD equipped with impedance monitoring and who are known with chronic heart failure of any cause
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
clinical efficacy and value of ambulatory intrathoracic impedance measurement of the Optivol alert as an indicator of decompensated heart failure reflected by sensitivity and positive predictive value | end of follow-up

SECONDARY OUTCOMES:
influence of left ventricular filling pattern and brain natriuretic level on the positive predictive value of the Optivol alert | end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: P Houthuizen, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven; A Meijer, MD PhD, Study Director — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis, Eindhoven, Netherlands